CLINICAL TRIAL: NCT04351516
Title: Randomized Controlled Trial of Hydroxychloroquine Versus Placebo in Early Ambulatory Diagnosis and Treatment of Elderly COVID19 Patients
Brief Title: Test and Treat COVID 65plus+
Acronym: COVID65plus
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No Patients enrolled
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID65plus; 2020-001482-37 (EudraCT Number)
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV 2; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydroxychloroquine (Experimental)
  Interventions: Drug: Hydroxychloroquine
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — dose of 600mg on the first day followed with 400mg/day divided in 2x200mg for 6 more days
  Arms: hydroxychloroquine
Other: Placebo — Placebo: Film Coated Tablette
  Arms: Placebo

SUMMARY:
Patients over equal or older than 65 yearswill be treated with a hydroxychloroquine versus placebo reduced loading dose of 600mg on the first day followed with 400mg/day divided in 2x200mg for 6 more days resulting in a total duration of therapy of 7 days. Measurement of Hydroxychloroquine-levels will be performed on day 7, . A follow-up by video or telephone conference will be performed to observe drug intake and collect adverse events during treatment phase on a daily base on working days and once during the weekend (i.e. 6 out of 7 days). After treatment phase follow-up by telephone calls will be done on day 10, 30, 60 (+/- 2 days).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 65 years
* Mild to moderate symptomatic respiratory tract Infection defined as not requiring hospital admission: SpO2 >94%, respiratory rate <20, mental state alert, no signs of septic shock
* Proven SARS-Cov2 infection by throat swab (PCR)
* Onset of symptoms within the last 3 days before randomization
* Must be able to adhere to the study visit schedule and other protocol requirements in the investigator's opinion. I.e. must be able to answer to questions concerning symptoms and side effects and must be able to consent to the informed consent.

Exclusion Criteria:

* Hospitalization at study inclusion
* Weight <50 kg
* Acute myocardial infarction
* Severe heart failure, characterized as NYHA class 3 or 4
* Use of concomitant medications that prolong the QT/QTc interval.
* QTc >450ms
* Bilirubin ≥ 1,5 x UNL, (except for known M. Meulengracht)
* AST/ALT ≥ 3 x ULN
* Albumine ≤ 2.8 g/dl
* Hemoglobin ≤ 9 g/dl
* Leucocytes ≤ 2000/µl
* Neutrophiles ≤ 1000/µl
* Thrombocytes ≤ 100.000/µl
* Troponin elevation
* BNP > 500 pg/ml
* Creatine kinase > 5 x ULN
* Creatinine >1,5 mg/dl
* Uncorrected hypopotassemia or hypomagnesemia
* History of hypoglycemic events
* History of or present cardial arrhythmia (except atrial fibrillation or paroxysmal supraventricular tachycardia)
* Bradycardia < 60 beats/min
* History of Retinopathy or Maculopathy
* Psoriasis
* Myasthenia gravis
* Epilepsy
* Immunodeficiency syndromes or need for highly immunosuppressive medication
* Pre-existing medication with hydroxychloroquine
* Known G6PD deficiency.
* Participation in another interventional study
* Known hypersensibility to hydroxychloroquine and its derivates

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
● Rate of hospitalization or death at day 7 after study inclusion | 7 days

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Uniklinikum Tuebingen, Tübingen
  - Uniklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gopel S, Bethge W, Martus P, Kreth F, Iftner T, Joos S, Dobele S, Mordmuller B, Kremsner P, Ettrich T, Seufferlein T, Bitzer M, Malek N. Test and treat COVID 65 plus - Hydroxychloroquine versus placebo in early ambulatory diagnosis and treatment of older patients with COVID19: A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jul 10;21(1):635. doi: 10.1186/s13063-020-04556-z. PMID 32650818